CLINICAL TRIAL: NCT02880579
Title: Evaluation of Clinical Results of Treatment of Cerebral Artery Occlusion by Mechanical Thrombectomy, in the Acute Phase of Stroke
Brief Title: Neurothrombectomy France
Acronym: NTF
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC11_0097
Record Dates: First submitted 2016-08-05; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Cerebral Artery Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Ischemic Brain Vascular Accident (CVA) is a major public health issue. An Early and appropriate charging anyone with stroke is essential to reduce mortality, reduce dependency and promote recovery of autonomy. Intravenous fibrinolysis in patients with cerebral infarction (NINDS 1995), is reserved for a small proportion of highly selected patients. It therefore remains a significant therapeutic challenge, especially for patients with against-indications to fibrinolysis or in whom there is no immediate benefit. For twenty years of mechanical devices have been developed to remove, as quickly as possible, the cause of intracranial arterial occlusion and allow restoration of blood flow before brain damage is irreversible.

NTF The protocol is part of the evaluation process of our clinical practices recommended by the National Health Authority (HAS), in the specific context of mechanical thrombectomy performed in French centers of interventional neuroradiology working with neurovascular units (A V).

ELIGIBILITY:
Inclusion Criteria:

* Signature of the information notice by the patient or his legal representative
* Age> 18 years
* Clinical and imaging consistent with ischemic stroke whose symptoms start back within 8h
* Thrombosis (TICI 0 or 1) of the carotid T, M1, M1-M2 bifurcation of the basilar artery occlusion in TANDEM ACI / M1.

Exclusion Criteria:

* Pregnant or lactating women
* Rapid improvement of NIHSS (gain of more than 4 points) between two pre-treatment assessments.
* ASPECT score <7 on the scanner or <5 on the diffusion-weighted imaging (DWI)
* Intracranial hemorrhage on imaging
* Inability of clinical evaluations at 3 months
* extensive lesions of the brain stem (the presence of a complete section of the brainstem hyperintense b1000)
* 0 Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 consecutive patients admitted to a stroke unit for cerebral infarction treated by thrombectomy included (with or without fibrinolysis by intra venous) prospectively over a period of 1 year and 3 months followed for clinical neurological assessment (primary endpoint) .
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
clinical score for handicap (mRS) | at 3 months

SECONDARY OUTCOMES:
hemorrhagic complications on postoperative imaging | baseline
hemorrhagic complications on postoperative imaging | at 1 day
physiological parameter : age | baseline
  Factors of good clinical prognosis
presence of coronary artery disease | baseline
  Factors of good clinical prognosis
presence of arterial hypertension | baseline
  Factors of good clinical prognosis
presence of diabetes | baseline
  Factors of good clinical prognosis
presence of hypercholesterolemia | baseline
  Factors of good clinical prognosis
presence of intracranial stenosis | baseline
  Factors of good clinical prognosis
presence of occlusive arterial disease | baseline
  Factors of good clinical prognosis
presence of haematological disorders | baseline
  Factors of good clinical prognosis
presence of neoplasia | baseline
  Factors of good clinical prognosis
NIHSS score | baseline
  Factors of good clinical prognosis
ASPECTS score | baseline
  Factors of good clinical prognosis
MRI imaging of stroke | baseline
  Factors of good clinical prognosis
unblocking rate based on the score TICI | at 3 months
NIHSS evaluation | at 24h
Influence of collaterality score on the NIHSS | at 24h
Influence ASPECTS score on the NIHSS | at 24h
Influence ASPECTS score on the NIHSS | at 3months
influence of anesthesia on the NIHSS | at 24h
hemorrhagic complications | at 24h
Influence of hemorrhagic complications on NIHSS | at 24h
Influence of hemorrhagic complications on NIHSS | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hubert DESAL, PU-PH, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided